CLINICAL TRIAL: NCT00848900
Title: A Controlled Clinical Trial of the Effect of Increases Time Outdoors in the Prevention of Juvenile-onset Myopia in Chinese Children
Brief Title: Guangzhou Outdoor Activity Longitudinal Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Mingguang He, Zhongshan Ophthalmic Center, ZOC
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GOAL2009
Record Dates: First submitted 2009-02-19; First posted 2009-02-20 (Estimated); Last update posted 2010-11-22 (Estimated); Status verified 2010-10

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention)
- Outdoor activity (Experimental): Adding 1 hour outdoor time into school curricula
  Interventions: Behavioral: Outdoor activity

INTERVENTIONS:
Behavioral: Outdoor activity — Adding 1 hour outdoor time into school curricula
  Arms: Outdoor activity

SUMMARY:
The purpose of this study is to assess whether outdoor activities are effective in preventing the development and progression of juvenile-onset myopia in Chinese children.

DETAILED DESCRIPTION:
1. To determine if increased engagement in outdoor activities reduces the development and progression of myopia in Chinese school children.
2. To identify the risk factors associated with the development and progression of juvenile-onset myopia.
3. To characterize the interaction between refractive error and education.

ELIGIBILITY:
Inclusion Criteria:

* All the students in Grade 1

Exclusion Criteria:

* No

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2009-04; Primary Completion 2012-04 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Cycloplegic refraction | 1 year

SECONDARY OUTCOMES:
Visual acuity | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mingguang He, PhD, MD, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] He M, Xiang F, Zeng Y, Mai J, Chen Q, Zhang J, Smith W, Rose K, Morgan IG. Effect of Time Spent Outdoors at School on the Development of Myopia Among Children in China: A Randomized Clinical Trial. JAMA. 2015 Sep 15;314(11):1142-8. doi: 10.1001/jama.2015.10803. PMID 26372583
- [Derived] Zhou Z, Morgan IG, Chen Q, Jin L, He M, Congdon N. Disordered sleep and myopia risk among Chinese children. PLoS One. 2015 Mar 26;10(3):e0121796. doi: 10.1371/journal.pone.0121796. eCollection 2015. PMID 25811755